CLINICAL TRIAL: NCT00494221
Title: A Two Part Study in Japanese Patients With mCRC, Consisting of an Open-label Phase I Part to Assess the Safety and Tolerability of Cediranib (AZD2171) in Combination With FOLFOX Followed by a Phase II, Randomised, Double-blind, Parallel Group Study to Assess the Efficacy of Cediranib (AZD2171) in Combination With FOLFOX
Brief Title: A Phase I/II Study of Cediranib (AZD2171) in Japanese Metastatic Colorectal Cancer Patients in Combination With FOLFOX
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D8480C00039
Record Dates: First submitted 2007-06-27; First posted 2007-06-29 (Estimated); Results first posted 2012-06-05 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-02

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal cancer; Recentin; Metastatic Cancer; FOLFOX
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — cediranib; Folfox protocol; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- FOLFOX + Cediranib 20 mg (Active Comparator): FOLFOX + Cediranib 20 mg
  Interventions: Drug: AZD2171; Drug: FOLFOX (5-fluorouracil, Leucovorin, Oxaliplatin)
- FOLFOX + Cediranib 30 mg (Active Comparator): FOLFOX + Cediranib 30 mg
  Interventions: Drug: AZD2171; Drug: FOLFOX (5-fluorouracil, Leucovorin, Oxaliplatin)
- FOLFOX + Placebo Cediranib (Placebo Comparator): FOLFOX + Placebo Cediranib
  Interventions: Drug: FOLFOX (5-fluorouracil, Leucovorin, Oxaliplatin); Drug: Placebo Cediranib

INTERVENTIONS:
Drug: AZD2171 — oral tablet
  Other Names: cediranib; RECENTIN™
  Arms: FOLFOX + Cediranib 20 mg; FOLFOX + Cediranib 30 mg
Drug: FOLFOX (5-fluorouracil, Leucovorin, Oxaliplatin) — intravenous infusion
  Other Names: Eloxatin®; 5-FU; Leucovorin
Drug: Placebo Cediranib — oral tablet
  Arms: FOLFOX + Placebo Cediranib

SUMMARY:
This Study is in two parts, the first part is to make sure that combining a potential new treatment, cediranib (AZD2171), with a standard treatment (FOLFOX) for metastatic colorectal cancer is safe. Once this part is complete and it is decided that it is safe to continue the Study will the go on to look at the efficacy of the two drugs together. This will be done by studying two treatment options. One will be the standard treatment alone (FOLFOX) + dummy cediranib (AZD2171) tablets and the other will be the standard treatment (FOLFOX) + real cediranib (AZD2171) tablets. Using dummy tablets means the study is 'blinded' and that non-one can tell the difference between the two treatment groups. This kind of study design is done to try to avoid the chance that the results might be biased in some way. The overall aim of the second part of the study is to see if adding cediranib (AZD2171) to a standard treatment for Metastatic Colorectal Cancer (mCRC), in this case FOLFOX, gives better results. That is, it's better than giving standard treatment alone in helping to prevent progression of mCRC.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic colorectal cancer
* WHO performance status 0-1
* Life expectancy is 12 weeks or longer

Exclusion Criteria:

* Patient with uncontrolled brain metastases
* Patient with inappropriate laboratory tests values
* Patient with poorly controlled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2007-06; Primary Completion 2009-10 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Robertson, Study Director — AstraZeneca; Hideyuki Mishima, M.D., PhD, Principal Investigator — National Hospital Organization Osaka National Hospital; Xiaojin Shi, MD, Study Chair — AstraZeneca
Locations (2):
- Japan (2):
  - Research Site, Osaka
  - Research Site, Saitama

REFERENCES:
- See also: CSR-D8480C00039.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=421&filename=CSR-D8480C00039.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomised=ITT=Safety: Cediranib 20mg=58, Cediranib 30mg=56, Placebo=58
Pre-assignment Details: PFS & OS: median based on Kaplan Meier analysis (i.e. adjusted for censored observations) but full range based on raw data (i.e. not adjusted for censored observations). OS: median non-estimable due to censored observations
Groups:
- Cediranib 20 mg: FOLFOX + Cediranib 20 mg
- Cediranib 30 mg: FOLFOX + Cediranib 30 mg
- Placebo: FOLFOX + Placebo
Period: Overall Study
Arm/Group | Cediranib 20 mg | Cediranib 30 mg | Placebo
Started | 58 | 56 | 58
Completed | 42 | 45 | 44
Not Completed | 16 | 11 | 14
Not completed — Death | 15 | 9 | 14
Not completed — Withdrawal by Subject | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cediranib 20 mg | Cediranib 30 mg | Placebo | Total
Number analyzed (Participants) | 58 | 56 | 58 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at informed consent
  years | 62.4 (9.3) | 62.1 (9.9) | 62.2 (9.6) | 62.2 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender at informed consent
  Participants
    Female | 20 | 26 | 19 | 65
    Male | 38 | 30 | 39 | 107

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Number of months from randomisation until progressive disease based on RECIST (progression of target lesions, clear progression of existing non-target lesions or the appearance of one or more new lesions) or death in the absence of progression.
Time Frame: RECIST at Baseline, Weeks 6, 12, 18, 24 and then every 12 weeks until progression through to a cut-off date of 13th Oct 2009 (based on approx 105 progression events observed across the 3 groups)
Measure: Median (Full Range); unit: Months
Arm/Group | Cediranib 20 mg | Cediranib 30 mg | Placebo
Number analyzed (Participants) | 58 | 56 | 58
Months | 10.23 [1.15 to 19.51] | 8.85 [0 to 19.47] | 8.32 [0.99 to 19.14]

2. Secondary Outcome: Objective Tumour Response Rate
Description: Number of patients with complete (CR) /partial response (PR) (based on RECIST). CR is defined as Disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of Longest Diameter (LD) of target lesions taking as reference the baseline sum LD.
Time Frame: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Cediranib 20 mg | Cediranib 30 mg | Placebo
Number analyzed (Participants) | 58 | 56 | 58
Participants | 31 | 39 | 31

3. Secondary Outcome: Best Percentage Change in Tumour Size
Description: Best percentage change in tumour size from baseline, based on the sum of the longest diameters of the target lesions
Time Frame: Randomisation until cut-off date 13OCT2009 (based on approximately 105 progression events observed across the 3 groups)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Cediranib 20 mg | Cediranib 30 mg | Placebo
Number analyzed (Participants) | 58 | 54 | 57
Percentage | -36.56 (24.52) | -43.99 (22.62) | -40.22 (35.84)

4. Secondary Outcome: Duration of Response
Description: Number of months from Complete/Partial response until progression up to cut-off date 13OCT2009 (based on approximately 105 progression events observed across the 3 groups).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Cediranib 20 mg | Cediranib 30 mg | Placebo
Number analyzed (Participants) | 31 | 39 | 31
Months | 13.26 (16.81) | 8.12 (6.18) | 10.42 (10.97)

5. Secondary Outcome: Overall Survival
Description: Number of months until death (censored if still alive at date cut-off). Median non-estimable if >50% of subjects within a group are censored.
Time Frame: Randomisation until cut-off date 13OCT2009 (based on approximately 105 progression events observed across the 3 groups)
Measure: Median (Full Range); unit: Months
Arm/Group | Cediranib 20 mg | Cediranib 30 mg | Placebo
Number analyzed (Participants) | 58 | 56 | 58
Months | NA [5.33 to 20.69] — Median non-estimable because >50% of participants were censored | 20.07 [0.59 to 20.53] | 19.51 [1.32 to 20.92]

ADVERSE EVENTS:
Groups:
- Cediranib 20 mg: Cediranib 20 mg
- Cediranib 30 mg: Cediranib 30 mg
- Placebo: Placebo
Arm/Group | Cediranib 20 mg | Cediranib 30 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 23/58 | 22/56 | 11/58
Other Adverse Events (participants affected / at risk) | 58/58 | 56/56 | 58/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cediranib 20 mg (N=58) | Cediranib 30 mg (N=56) | Placebo (N=58)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Cardiac Failure (Cardiac disorders) | 0 | 1 | 0
Prinzmetal Angina (Cardiac disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 2 | 0 | 4
Nausea (Gastrointestinal disorders) | 4 | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 0
Anal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal Perforation (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 1 | 0
Mesenteric Artery Thrombosis (Gastrointestinal disorders) | 0 | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 3 | 0 | 0
Fatigue (General disorders) | 2 | 2 | 0
Malaise (General disorders) | 0 | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Anaphylactic Shock (Immune system disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1 | 0
Abdominal Abscess (Infections and infestations) | 0 | 0 | 1
Catheter Site Infection (Infections and infestations) | 0 | 1 | 0
Wound Infection (Infections and infestations) | 0 | 1 | 0
Postoperative Ileus (Injury, poisoning and procedural complications) | 1 | 0 | 0
Weight Decreased (Investigations) | 2 | 0 | 0
Blood Creatinine Increased (Investigations) | 1 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 10 | 5 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bile Duct Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Altered State Of Consciousness (Nervous system disorders) | 0 | 1 | 0
Brain Stem Infarction (Nervous system disorders) | 1 | 0 | 0
Cerebral Haemorrhage (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 0 | 1
Reversible Posterior Leukoencephalopathy Syndrome (Nervous system disorders) | 0 | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0 | 0
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cediranib 20 mg (N=58) | Cediranib 30 mg (N=56) | Placebo (N=58)
Anaemia (Blood and lymphatic system disorders) | 6 | 7 | 3
Neutropenia (Blood and lymphatic system disorders) | 6 | 3 | 1
Hypothyroidism (Endocrine disorders) | 5 | 6 | 1
Diarrhoea (Gastrointestinal disorders) | 52 | 48 | 22
Nausea (Gastrointestinal disorders) | 37 | 36 | 37
Stomatitis (Gastrointestinal disorders) | 32 | 29 | 25
Vomiting (Gastrointestinal disorders) | 23 | 27 | 14
Constipation (Gastrointestinal disorders) | 21 | 14 | 15
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 4 | 8
Haemorrhoids (Gastrointestinal disorders) | 6 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 3 | 5 | 4
Cheilitis (Gastrointestinal disorders) | 5 | 3 | 4
Gingivitis (Gastrointestinal disorders) | 5 | 5 | 1
Dental Caries (Gastrointestinal disorders) | 4 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 4
Periodontitis (Gastrointestinal disorders) | 4 | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 3 | 0
Anal Haemorrhage (Gastrointestinal disorders) | 2 | 3 | 1
Ascites (Gastrointestinal disorders) | 3 | 1 | 0
Glossitis (Gastrointestinal disorders) | 3 | 1 | 1
Toothache (Gastrointestinal disorders) | 3 | 1 | 2
Fatigue (General disorders) | 38 | 40 | 36
Pyrexia (General disorders) | 8 | 12 | 11
Oedema Peripheral (General disorders) | 5 | 7 | 2
Influenza Like Illness (General disorders) | 4 | 3 | 5
Mucosal Inflammation (General disorders) | 3 | 1 | 1
Hepatic Function Abnormal (Hepatobiliary disorders) | 3 | 3 | 0
Drug Hypersensitivity (Immune system disorders) | 6 | 9 | 12
Nasopharyngitis (Infections and infestations) | 14 | 10 | 6
Oral Candidiasis (Infections and infestations) | 4 | 1 | 0
Cystitis (Infections and infestations) | 3 | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 38 | 42 | 38
Dehydration (Metabolism and nutrition disorders) | 3 | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 11 | 5 | 5
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 1
Neuropathy Peripheral (Nervous system disorders) | 42 | 35 | 38
Dysgeusia (Nervous system disorders) | 18 | 17 | 18
Peripheral Sensory Neuropathy (Nervous system disorders) | 7 | 15 | 11
Headache (Nervous system disorders) | 6 | 6 | 6
Insomnia (Psychiatric disorders) | 4 | 2 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 24 | 16 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15 | 19 | 9
Hiccups (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 6
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 31 | 34 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 12 | 17 | 15
Rash (Skin and subcutaneous tissue disorders) | 12 | 12 | 8
Pigmentation Disorder (Skin and subcutaneous tissue disorders) | 8 | 5 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 3 | 7
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 | 7 | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 5 | 2 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 5 | 0 | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 4 | 4 | 1
Haemorrhage Subcutaneous (Skin and subcutaneous tissue disorders) | 4 | 2 | 0
Hypertension (Vascular disorders) | 47 | 47 | 18
Hypotension (Vascular disorders) | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a Study Site, or an investigator, requests permission to publish data from this study, any such publication (including oral presentations) is to be agreed with AstraZeneca prior to publication.